CLINICAL TRIAL: NCT04137497
Title: Behavioral Assessment of Nociception on the Nociception Coma Scale-Revised in Patients With Disorders of Consciousness: A Sign of Consciousness
Brief Title: Behavioral Assessment of Nociception on NCS-R
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Other Study IDs: 2017N54965
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Disorder of Consciousness; Unresponsive Wakefulness Syndrome; Minimally Conscious State
Keywords: disorders of consciousness; unresponsive wakefulness syndrome; minimally conscious state; Nociception Coma Scale-Revised
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with disorders of consciousness
  Interventions: Diagnostic Test: The Coma Recovery Scale-Revised and the Nociception Coma Scale-Revised (NCS-R)
- Patients with unresponsive wakefulness syndrome
  Interventions: Diagnostic Test: The Coma Recovery Scale-Revised and the Nociception Coma Scale-Revised (NCS-R)
- Patients with minimally conscious state
  Interventions: Diagnostic Test: The Coma Recovery Scale-Revised and the Nociception Coma Scale-Revised (NCS-R)

INTERVENTIONS:
Diagnostic Test: The Coma Recovery Scale-Revised and the Nociception Coma Scale-Revised (NCS-R) — All enrolled DOC patients were evaluated at least five times over one week by two trained professionals using the Chinese version of the CRS-R. During the evaluation of the patient's consciousness level, the NCS-R was used to evaluate the pain response of all patients in random order at least once, and the best behavioral response (i.e., the highest score) of each subscale was recorded during resting, noxious, and physiotherapy conditions, respectively, according to the NCS-R guidelines.

SUMMARY:
The aim of this study was to investigate the relationship between behaviorally assessed consciousness levels and responsiveness to nociception in patients with disorders of consciousness (DOC)

DETAILED DESCRIPTION:
Patients with a clinical consensus of DOC were enrolled. The Coma Recovery Scale-Revised (CRS-R) was used to assess the DOC patients' consciousness levels and the Nociception Coma Scale-Revised (NCS-R) was used to evaluate their pain response over one week. Furthermore, the relationship between behaviorally assessed consciousness levels and pain response was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* (1) at least 18 years old
* (2) acquired brain injury
* (3) no neuromuscular blockers or sedatives used within 72 hours of enrollment.

Exclusion Criteria:

* (1) functional disorders caused by progressive mental diseases
* (2) persistent seizures
* (3) unstable vital signs
* and/or (4) double upper-limb frustration, fracture.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All enrolled DOC patients were evaluated at least five times over one week by two trained professionals using the Chinese version of the CRS-R. The highest score was selected as the final bedside behavioral diagnosis of the patient's consciousness level. During the evaluation of the patient's consciousness level, the NCS-R was used to evaluate the pain response of all patients in random order at least once, and the best behavioral response (i.e., the highest score) of each subscale was recorded during resting, noxious, and physiotherapy conditions, respectively, according to the NCS-R guidelines. The patient's specific behavioral performance was also recorded.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
Nociception Coma Scale-Revised | Within 7 days
  The Nociception Coma Scale-Revised was used to evaluate the pain response of all patients in random order at least once. A score greater than or equal to 3 points indicated that the patient was responsive to pain stimulation, while a score greater than or equal to 4 points suggested that the patient might have pain perception related to consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro., Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Schnakers C, Chatelle C, Vanhaudenhuyse A, Majerus S, Ledoux D, Boly M, Bruno MA, Boveroux P, Demertzi A, Moonen G, Laureys S. The Nociception Coma Scale: a new tool to assess nociception in disorders of consciousness. Pain. 2010 Feb;148(2):215-219. doi: 10.1016/j.pain.2009.09.028. Epub 2009 Oct 24. PMID 19854576
- [Background] Chatelle C, Majerus S, Whyte J, Laureys S, Schnakers C. A sensitive scale to assess nociceptive pain in patients with disorders of consciousness. J Neurol Neurosurg Psychiatry. 2012 Dec;83(12):1233-7. doi: 10.1136/jnnp-2012-302987. Epub 2012 Aug 20. PMID 22906615
- [Background] Sattin D, Pagani M, Covelli V, Giovannetti AM, Leonardi M. The Italian version of the Nociception Coma Scale. Int J Rehabil Res. 2013 Jun;36(2):182-6. doi: 10.1097/MRR.0b013e3283618d68. PMID 23603804
- [Background] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Comprehensive Systematic Review Update Summary: Disorders of Consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Arch Phys Med Rehabil. 2018 Sep;99(9):1710-1719. doi: 10.1016/j.apmr.2018.07.002. Epub 2018 Aug 8. PMID 30098792